CLINICAL TRIAL: NCT04148963
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Efficacy and Safety Study of Staccato Loxapine (ADASUVE®) for Inhalation in Acutely Agitated Patients With Schizophrenia or Bipolar Disorder
Brief Title: A Study of Staccato Loxapine (ADASUVE®) for Inhalation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADS-ZK-2019
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-01

CONDITIONS: Psychomotor Agitation; Schizophrenia; Bipolar Disorder
Keywords: schizophrenia; bipolar disorder; agitation; inhaled loxapine; ADASUVE
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia; Bipolar Disorder | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled loxapine (Experimental): Inhaled Loxapine 9.1 mg, may repeat x 1 or 2 after 2 hours
  Interventions: Drug: Inhaled loxapine
- Inhaled placebo (Placebo Comparator): Inhaled placebo, may repeat x 1 or 2 after 2 hours
  Interventions: Drug: Inhaled placebo

INTERVENTIONS:
Drug: Inhaled loxapine — Inhaled Loxapine 9.1 mg, may repeat x 1 or 2 after 2 hours
  Other Names: ADASUVE
  Arms: Inhaled loxapine
Drug: Inhaled placebo — Inhaled placebo, may repeat x 1 or 2 after 2 hours
  Arms: Inhaled placebo

SUMMARY:
Phase 3 safety and efficacy study of Staccato Loxapine in the treatment of acute agitation in schizophrenic or bipolar disorder patients.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel group, efficacy and safety study of Staccato Loxapine or placebo in treating acute agitation in patients with schizophrenia or bipolar disorder (manic or mixed episodes) as defined by DSM-V criteria.Patients may receive up to 3 doses of study drug in a 24-hour period, depending on their clinical status. The primary endpoint is the change from baseline in the PANSS (Positive and Negative Symptom Scale) Excited Component (also known as PEC) score, performed at 2 hours after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female patients between the ages of 18 to 65 years, inclusive.
* 2. Patients who met Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for schizophrenia or bipolar disorder.
* 3. Patients are judged to be clinical mild to moderate agitation at baseline with a total value of ≥ 14, and have a score ≥4 on at least 1 of 5 items on the PANSS-EC scale, and with a value of ≥3 on CGI-S scale.
* 4. Patients are judged to be cooperative by the Investigator.
* 5. Written informed consent from patients (and/or legally acceptable representative, legally acceptable representative preferred) is obtained.

Exclusion Criteria:

* 1. Patients with agitation caused primarily by Delirium, Dpilepsy, Developmental Retardation, acute alcohol or psychoactive drugs intoxication/withdrawal symptoms (as per Investigator's judgment).
* 2. Patients judged to be at serious risk for suicide as per the Investigator's judgement.
* 3. Patients with a history of allergy or intolerance to loxapine or amoxapine.
* 4. Female patients of childbearing potential who have a positive urine pregnancy test at screening or breastfeeding.
* 5. Patients with acute respiratory signs/symptoms (e.g., wheezing) or with active airways disease (such as patients with asthma or chronic obstructive pulmonary disease).
* 6. Patients who are considered by the Investigator, for any reason, to be unsuitable candidates for receiving inhaled loxapine, or are likely to be unable to use the inhalation device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in PANSS-EC From Baseline | Time Frame: Baseline and 2 hours
  The Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (min) to 7 (max). The PANSS-EC, the sum of these 5 subscales, thus ranges from 5 to 35. Individuals were eligible if they had a PANSS-EC of ≥14 (out of 35) and a score ≥4 (out of 7) on at least 1 of the 5 items.

SECONDARY OUTCOMES:
Change in PANSS-EC From Baseline | Baseline and 30 minutes
Change in PANSS-EC From Baseline | Baseline and 4 hours
Change in PANSS-EC From Baseline | Baseline and 24 hours